CLINICAL TRIAL: NCT06555107
Title: Acute Preoperative Pain and Chronic Post-surgical Pain in Emergency Surgery
Acronym: POCSE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2024_843_0038
Record Dates: First submitted 2024-08-13; First posted 2024-08-15 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Chronic Postsurgical Pain; Acute Pain; Emergency Surgery; Opioid; Postoperative Pain; Risk Factors
Keywords: risk factors; Chronic Postsurgical Pain; Acute Pain; emergency surgery; opioid; Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative; Acute Pain | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaire — Patients included in the study will be asked to complete a questionnaire 48 to 72 hours after surgery to assess their perception of pain and preoperative anxiety
Other: phone call — Patients will then be interviewed by phone 3 months after their emergency surgery. During the interview, they will be questioned via a standardised questionnaire on the existence of CPSP

SUMMARY:
Studies evaluating postoperative pain as a risk factor for CPSP are almost exclusively carried out in the context of scheduled surgery. As a result, the preoperative pain studied as a risk factor for chronicity is essentially a state of pain that has persisted for several weeks or even several months.

In emergency surgeries, patients are subject to acute preoperative pain of varying intensity and the duration of which may vary by a few days. A few studies have highlighted the intensity of acute preoperative pain as a factor favouring moderate to severe postoperative pain. At this point, no study has addressed the long-term consequences of this intense preoperative pain the emergency context.

An evaluation in the field of emergency surgery, where the preoperative pain is often intense and limited in time, would enable us to identify more precisely the impact of acute pain on the incidence of CPSP.

The investigators are hypothesising that the occurrence of CPSP at 3 months in patients undergoing emergency orthopaedic or abdominal surgery is associated with acute preoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old.
* Emergency orthopaedic and/or abdominal surgery.
* Informed consent.
* Affiliation to a social security scheme

Exclusion Criteria:

* Intraoperative complications that are life-threatening or require the surgical procedure to be discontinued.
* Post-operative intensive care unit admission.
* Ambulatory surgery.
* Endoscopic surgery.
* Repeat surgery at the same site in less that 3months.
* Pregnant or breast-feeding patients.
* Patients under guardianship or deprived of liberty.
* Patients suffering from psychiatric pathologies.
* Patients suffering from neurodegenerative pathologies.
* Patients for whom self-assessment of pain using a numerical scale (0-10) cannot be carried out (non-communicative patients, non-French-speaking patients, and so on).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 693 (Estimated)
Dates: Start 2024-08-29 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Frequency of CPSP | at 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens-Picardie, Amiens, France

IPD SHARING:
Plan to Share IPD: No